CLINICAL TRIAL: NCT00936689
Title: Treatment of Hepatocellular Carcinoma (HCC)by Selective Traditional Chemoembolization(TACE)Versus Selective TACE Via Microspheres Loaded With Doxorubicin: a Multicentre,Randomized,Open Label,Controlled Study.
Brief Title: Traditional (Traditional Chemoembolization) TACE Versus Microsphere TACE
Acronym: PRECISION-IT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rita Golfieri (Other)
Responsible Party: Sponsor-Investigator, Rita Golfieri, MD, University of Bologna
Organization: University of Bologna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAD01; EudraCT 2006-003034-15
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma;; Chemoembolization;; DC-Beads.
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional TACE (Sham Comparator): Chemoembolization by standard technique: epirubicin (maximum dose of 75 mg) conjugated with an oil-based contrast medium (Lipiodol) at the maximum dose of 15 ml + gelatin sponge particles(particles of transient embolization material, required to obstruct the treated vessel).
  Interventions: Procedure: Selective traditional TACE
- TACE with microsphere (Active Comparator)
  Interventions: Procedure: Selective TACE via microsphere loaded with Doxorubicin

INTERVENTIONS:
Procedure: Selective TACE via microsphere loaded with Doxorubicin — Chemoembolization with microspheres: doxorubicin (maximum dose of 75 mg x vials of microspheres) loaded with non-reabsorbable microspheres (sulfate hydrospheres) at the dose of 2 ml per vial (definitive embolization).
  Other Names: DC-beads
  Arms: TACE with microsphere
Procedure: Selective traditional TACE — Traditional chemoembolization: epirubicin (maximum dose of 75 mg) conjugated with Lipiodol at the maximum dose of 15 ml + Spongel.
  Other Names: TACE
  Arms: Traditional TACE

SUMMARY:
Background

Hepatic intra-arterial chemoembolization (TACE) is proposed when potentially curative therapy (eg. surgical resection, percutaneous ablation)is no longer possible. Prospective and non-randomized retrospective studies showed TACE to be capable to increase survival vs controls. In 2002 the first results of two RCTs were published which had been conducted on unresectable HCC patients, designed to assess the impact produced by TACE on survival, demonstrated a statistically significant advantage in TACE treated patients compared to controls. The same results have been confirmed by a meta-analysis conducted on 14 trials published in literature. The limitations of TACE are represented however by the difficulties in obtaining a complete necrosis of the lesion treated and for this reason new embolization agents are being developed to increase the efficacy of TACE in HCC as the microsphere, in poly vinyl alcohol and co-acrylic acid that are not reabsorbable and induce permanent embolization. The first experimental studies using microsphere showed the good tolerability and the higher rate of tumor necrosis, but no RCTs have been conducted to investigate their impact on survival. Objectives. The primary aim of this study is to compare 2 years survival of patients randomized to selective traditional TACE or selective TACE via microspheres loaded with Doxorubicin. Secondary objectives investigate the time to progression of disease (radiologic and symptomatic) by radiologic, laboratory tests and the QoL questionnaire administration. Methods. This is a multicentre, randomized, open-label, active controlled study in HCC patients treated with standard TACE vs TACE with doxorubicin - loaded microsphere. The study comprises a selection period, a treatment period and a follow up phase with a total duration of 2 years from randomization. Expected results. The sample size(alfa 5%, power 80%) is adequate to detect a 20% difference between TACE with microsphere vs traditional TACE.

DETAILED DESCRIPTION:
INTRODUCTION

Hepatocellular carcinoma (HCC) is one of the most frequent malignancies in man. Liver transplantation, surgical resection and percutaneous ablation (alcoholization and thermal ablation) are curative therapies and can be used only in patients presenting with early phase disease, whereas 50-70% of HCC diagnoses are made when the disease has already reached the intermediate-advanced phase.

For HCC for which potentially curative therapy is no longer possible, palliative treatment has been proposed by hepatic intra-arterial chemoembolization (TACE) consisting of an infusion of cisplatin or doxorubicin emulsified with lipiodol, followed by a transient flow blockage achieved by reabsorbable particles (gelatin sponge particles). The rationale for the intra-arterial administration of chemotherapy agents in association with embolization material lies in the presence of double hepatic vascularization: hepatocytes are mainly vascularized by the portal structure (approximately 90%) whereas malignant cells are vascularized by the arterial structure (approximately 90%).

Prospective and non-randomized retrospective studies showed TACE to be capable of increasing survival (60-88% at one year, 30-60% at 2 years and 18-50% at 3 years) versus controls.

Despite these encouraging results, none of the first six RCT studies investigating TACE showed a significant increase of survival but only a decrease in tumor dimension. These trials however included mainly large tumors, in patients with severe liver disease, and these conditions may well have masked the benefits offered by TACE.

In 2002 the first results of two RCTs were published which had been conducted on unresectable HCC patients, designed to assess the impact producted by TACE on survival, and which demonstrated a statistically significant advantage in TACE-treated patients compared to controls: survival at 1, 2, and 3 years was 82%, 63%, and 29%, respectively, in the TACE arm versus 63%, 27%, and 17%, respectively, in the control group of the Llovet study, and survival at 1, 2, and 3 years was 57%, 31%, and 26%, respectively, in the TACE arm versus 32%, 11%, and 3%, respectively, the control group of the study conducted by Lo. Both studies confirmed that TACE was a safe procedure, with a low complication rate and that incidence of liver failure had not increased by a significant percentage in the TACE-treated group. A recent, systematic meta-analysis conducted on 14 trials published in literature, appropriately chosen to compare effects on survival exerted by TACE compared to the conservative treatment with tamoxifen confirmed the aforesaid findings.

The limitations of TACE are represented however by the difficulties in obtaining a complete necrosis of the lesions treated, and for this reason new embolization agents are being developed to increase the therapeutic efficacy of chemoembolization in HCC.

Such newly developed materials include the increasingly interesting expansible, high biocompatibility microspheres in poly(vinyl alcohol and co-acrylic acid) with the following novel features capable of enhancing anticancer effects: 1) they are not reabsorbable, and induce permanent embolization; 2) being deformable they adapt to the morphology of the vessels to be embolized, and selectively target cancerous arterial capillaries: 3) they deliver greater quantities of chemotherapy agent, minimizing systemic effects thereof.

The first experimental studies on the use of microspheres in HCC patients showed that such therapy is well tolerated and causes a higher rate of necrosis compared to standard TACE, but as of today, no RCTs have been conducted to investigate their impact on survival.

STUDY PLAN

- Study design: This is a multicentre, randomized, open-label, active-controlled study in HCC patients treated with standard chemoembolization versus chemoembolization with doxorubicin-loaded microspheres. The study comprises a selection phase, a treatment period and a follow-up period, with a total duration of 2 years from randomization.

During the screening phase laboratory tests and diagnostic imagings (Ultrasound/CAT scan/MRI) will be performed (as indicated in the inclusion criteria).

- Study population: The study population will be composed of 214 inpatients presenting with HCC, 107 per each randomization arm.

TREATMENTS

- Study treatments: Both arms will receive chemotherapy (epirubicin or doxorubicin) via hepatic intra-arterial delivery + intra-arterial chemoembolization of the study arterial branches to be treated

Arm A: chemoembolization by standard technique: epirubicin (maximum dose of 75 mg) conjugated with an oil-based contrast medium (Lipiodol) at the maximum dose of 15 ml + gelatin sponge particles (particles of transient embolization material, required to obstruct the treated vessel)

Arm B: chemoembolization with microspheres: doxorubicin (maximum dose of 75 mg x vials of microspheres) loaded with non-reabsorbable microspheres (sulfate hydrospheres) at the dose of 2 ml per vial (definitive embolization). The chemotherapy agent is released over a 14-day period, with a concentration peak in the tumor at 72 hours from treatment, and tumor concentration which is 100-fold that achieved by traditional intra-arterial injection. Half life of the drug is about 10 times longer than traditional TACE, with a systemic concentration of the drug which is 100 times less than that observed with standard TACE.

As a rule the procedure is performed once per each HCC lesion treated, since the microspheres exert definitive chemoembolization action; any repeated treatment on the same nodule is possible only whem the presence of partial persistence of vascularization is observed during the imaging assessment during follow-up.

- Assignment to treatment: At visit 1, a unique alphanumeric identification code will be assigned to eligible patients. Codes which have been assigned to patient who then discontinue participation cannot be thereafter reassigned.

Patients who meet inclusion and exclusion criteria will be randomized to one of two study treatments. Patient assignment to treatment is performed based on the randomization list, and by allocating the first and lowest randomization code available. The randomization list will be generated by the Pharmacy - Investigational Drug Service - of the coordinating center and the relevant part thereof will be sent to the investigational sites The information relating to the randomization list are is strictly confidential and may be accessed only by authorized persons and the data concerning the study will be entered into the database at the time of the follow-up visits. An interim assessment of global survival is foreseen to occur once 50% of patients and the data relating to their first follow-up visit have been included into the database.

- Discontinuation of treatment: Each patient fully maintains the right to discontinue his/her participation in the study at any given time; moreover, should it be considered to be of benefit for his/her health, he/she may be withdrawn from the study by the physicians in charge of the study.

- Visits and assessment: The monthly visits (V1, V2 and V3) may be postponed by 7 days. The three-monthly visits (V4 and Vn) may be brought forward/postponed by 10 days.

- Selection visit: Before initiating any study specific procedure, the investigator must obtain the written informed consent from the patient, Screening evaluations include laboratory tests, a physical examination, a pregnancy test for women of childbearing potential. In case results should be available for such exams which were performed within one month previously they do not have to be repeated. Evaluations will be recorded in the CRF at the Visit 1 page only if the patient is eligible.

Laboratory tests:

1. Creatinine 2. Bilirubin 3. GPT 4. Albumin 5. Hemoglobin 6. WBC 7. PLT 8. PT

EFFICACY EVALUATIONS

Efficacy of the treatment will be assessed at V3 and at V4 and Vn by means of the following:

1. visit and completion of the attached questionnaires, or in case the patient cannot come for the visit, by means of a telephone interview
2. the above-listed laboratory tests to assess evaluation of the disease
3. abdominal CAT scan or MRi to asses radiological evaluation of the disease
4. α-fetoprotein to assess biohumoral levels of the disease

   SAFETY EVALUATIONS

   Evaluation of safety of the treatment will consist in monitoring and recording adverse events, serious adverse events, laboratory tests and measurement of vital signs.
   * Adverse events:

   Information relating to all of the adverse events, those reported spontaneously by the subject and those identified by the Investigator pursuant to specific questions, as well as those identified through the physical examination of the patient, laboratory tests or other, will be collected, recorded on the CRF and followed as appropriate.

   - Serious Adverse Events: Information concerning all serious adverse events will be collected and recorded on the Serious Adverse Event reporting form. So as to guarantee patient safety, all serious adverse events must be notified to the Ethics Committee within 24 hours from the time they have come to the knowledge of the Investigator, by means of the specific SAE form.
   * Contact persons:

   Adverse events must be reported to the Principal Investigator and notified to the Ethics Committee Telephone and fax numbers of the contact persons for notification of Serious Adverse Events and Pregnancies are listed in the 'Investigator Folder provided to each site.

   DATA MANAGEMENT AND STATISTICAL ANALYSIS

   - Data management: Personnel appointed by the Investigator must record the information required by the protocol on the Case Report Form (CRF).

   The data contained in the CRF will be data entered centrally by personnel appointed thereto by the Clinical Principal Investigator by single data entry and electronic verification of data. Any text elements (eg, comments) will be verified manually. Data entries will subsequently be controlled by validation programs and listing controls. Obvious errors will be corrected directly by data management personnel, other errors or omissions will instead be recorded on Data Query forms which will be sent to the Investigators for resolution.

   Information relating to concomitant treatments will be codified based on the WHO Drug Reference List, which makes use of the Anatomic Therapeutic Chemical (ATC) classification. Concomitant diseases and adverse events will be codified using the ICD9 classification terminology.

   The database will be closed once it has been confirmed to be complete and accurate. Any changes made to the data after database lock may be performed solely if agreed to in writing by the Principal Investigator, the Statistician, the authors of the protocol and the collaborators appointed thereby to complete CRF and the database.

   - Statistical methods: This study intends to assess efficacy and tolerability of chemoembolization with microspheres versus chemoembolization by standard technique. The data collected will be grouped and summarized against demographic variables, baseline characteristics and efficacy and safety assessment. Exploratory analyses will be carried out using descriptive statistics. The data will be presented both on the "intent-to-treat" population (in other words, all the patients who have completed the study without any major protocol violations, such as for instance performance of alternative treatments for hepatocarcinoma or unjustified refusal to continue the study and undergo monitoring).

   An interim evaluation to assess overall survival will be carried out once 50% of the patients foreseen have been enrolled and the data relating to the first follow-up visit have been entered into the database.

   Safety evaluations will be based mainly on the frequency of adverse events, including all of the serious adverse events. Adverse events will be summarized presenting per each treatment group the number and percentage of patients who have presented any adverse event whatever, an adverse event in a specific body system and a specific adverse event. Any other information collected (i.e., the severity or correlation with the study drug) will be codified as appropriate.

   Moreover, analytical lists will be drafted illustrating details concerning:

<!-- -->

1. patients who have discontinued the study and correlated reasons:
2. patients who have discontinued the study due to adverse events;
3. patients who have experienced serious adverse events.

   * Characteristics of data sets, treatments and concomitant diseases:

   Data relating to demographics and baseline characteristics, and regarding efficacy and safety observations and parameters will be summarized, as will likewise be done for the main concomitant diseases recorded upon inclusion into the study. Listings will be created for patients who discontinue the study and will describe the reasons therefore.

   - Efficacy evaluation: Primary variable The primary efficacy evaluation will be carried out on the ITT population (intention to treat) comprised of all randomized patients.

   The primary efficacy variable is represented by survival at Month 24 (favorable event). According the the ITT protocol, mortality by Month 24 and withdrawal from the study will be considered to be unfavorable events.

   Frequency of events will be recorded for both treatment groups and the comparison will be carried out by means of Fisher's exact test. Evaluation will be performed of the primary endpoint stratified per sex, age (median value), Child-Pugh class (A, B), alpha-fetoprotein (median values).

   - Efficacy evaluation: Secondary variables Secondary efficacy variables will be assessed both as per ITT (intent to treat population) and PPP (per protocol population) procedures.

   Secondary variables will be described using: frequencies, mean values, standard deviations, 95% confidence intervals (95% CI), ranges and interquartile intervals in accordance with the type of variable taken into consideration.

   Continuous secondary variables will be assessed by means of variance analysis (ANOVA) using designs which are appropriate for the investigational protocol (by repeated measures for between-subject factors, two-way classification in case of stratified analyses, etc.) An estimate of effects assessed will also recorded.

   The secondary ordinal or nominal variables will be analyzed by non-parametric methods (Mann-Whitney, Wilcoxon, Fisher, McNemar, chi-squared tests, and by Mantel-Haenszel linear association).

   Finally, univariate and multivariate procedures will be applied by logistic analyses to assess both the effect of any interactions and to determine independence of significant factors detected by prior analyses.

   Statistical evaluations will be carried out by SPSS (Statistical Package for the Social Sciences: version 13.0 for Windows). Two-tailed probability value with three significant digits will be computed; any values below 0.05 will be considered statistically significant.

   - Safety evaluation: The safety analysis will be performed on the "Safety population", comprised of all patients included into the study and receiving chemoembolization.

   Adverse events will be summarized indicating number and percentage of patients with all types of events, classified per body system and per preferred term. The other information collected (eg. severity, causal correlation) will be listed as well as patients experiencing serious adverse events.

   Moreover, a listing will be created of patients who have experienced adverse events and who have discontinued the study due to adverse events.

   Laboratory test values will be summarized in appropriate tables showing frequency of values belong a predefined interval. Values representing relevant abnormalities will be listed.

   Other safety data (eg. electrocardiograms, vital signs and specific examinations) will be assessed as appropriate.

   - Sample size: The study was designed to demonstrate superiority of the effect of chemoembolization with microspheres versus standard chemoembolization on survival recorded 24 months after randomization (increase of survival by 20%).

   In particular, a 60% survival rate is expected in the chemoembolization with microspheres arm versus an expected survival rate of 40% in the group receiving standard treatment.

   It has been calculated that to detect a 20% difference between the two types of treatment, with an 80% power and a 5% significance level,a total number of 214 patients, 107 per treatment arm, must be enrolled.

   The sample size was calculated by the "Power calculator, UCLA Department of Statistics" software, applying Fisher's exact test.

   ADMINISTRATIVE PROCEDURES

   - Good Clinical Practice Rules: This study will be conducted in accordance with the Good Clinical Practice principles and of the declaration of Helsinki and in respect of national laws regulating conduction of clinical studies. By signing the protocol, the investigator agrees to comply with the procedures and instructions contained therein, and to conduct the study in conformity with GCP rules, the Declaration of Helsinki and national laws resulting clinical research.

   - Amendments to the protocol or any other change to study conduction: Any change to the protocol will be made in the form of an amendment. Any unforeseen change in study conduction will be recorded in the "Clinical Study Report".

   - Ethics committees and informed consent: The study protocol, any protocol amendment, the informed consent and any other information for patients must be approved by the Ethics Committee of the institution to which the Investigator is affiliated.

   As regards the amendments, the Investigator must immediately implement them after prior written communication to the Ethics Committee, and shall not await for the Ethics Committee to issue its approval whenever such amendment concerns the safety of patients taking part in the study. Moreover, should the Investigator believe that for reasons of patient safety it is necessary to immediately implement a change to the protocol, he/she must notify the Ethics Committee competent for the site within 10 work days.

   In order to take part in the study, each patient must release his/her written informed consent.

   - Archiving of documentation: The Investigator is responsible for archiving and storage of the essential documents of the study, prior to and throughout study conduction and after completion or interruption of the study itself, in accordance with and for the time period established by the provisions of existing applicable laws and by GCP rules.

   The data collected on the CRF will be rigorously anonymous and the subject will be identified solely by a number and his/her initials.

   The Investigator must store the original data of patients (for instance, demographics and medical information, laboratory data, electrocardiograms etc.) and a copy of the signed written informed consent. Prior to the initiation of the study, it may be established that certain data be recorded directly on the CRF, which in this case will be considered as a source document.

   - Inspections/Audits: The Principal Investigator or personnel appointed may perform verifications throughout the study to ensure that the study is being conducted in accordance with the protocol and with the provisions of existing applicable laws. Also Regulatory Authorities may conduct inspections on the study (both throughout its conduction or after completion of the study). Should a Regulatory Authority require an inspection, the Investigator must promptly notify the Ethics Committee thereof. By signing the protocol, the Investigator agrees to allows audits to be conducted both by appointed personnel and inspections by Regulatory Authorities.

   - Management of the investigational Medical Device: The investigational device (microspheres) will be provided by the Pharmacy in the marketed packages.

   The Investigator must ensure that it is used in conformity with the protocol. The Investigator and/or the pharmacist or another person competent therefore will be responsible for the storage of the product in a secure place, with limited access, maintaining in accordance with the storage conditions shown on the package.

   - Publication of results: Each formal presentation or publication of the data deriving from this study must be considered as a publication authored by the Investigator and by the professionals involved in the spontaneous study.

   - Privacy and Confidentiality: Documents pertaining to the study (eg. protocol, CRF and others) must be stored in a secure place to guarantee maintenance of confidentiality and privacy.

   - Study discontinuation: The party proposing the spontaneous study reserve the faculty to interrupt the study in case, throughout conduction thereof, and based on the results obtained by the interim analysis, conclusions should be reached not justifying the continuation of the study itself.

   - Contact persons: Telephone and fax numbers of the contact persons (i.e., the party proposing the spontaneous study and his/her collaborators) are listed in the 'Investigator Folder provided to each site.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HCC: based on the Guidelines issued by AASLD (American Association for the Study of Liver Diseases) (latest diagnostic radiological imaging performed within 1 month from enrolment)
* HCC for which transplantation, surgical resection or percutaneous ablation are not indicated
* Absence of extrahepatic cancer involvement
* Absence of portal vein thrombosis, with the exception of thrombosis of a segment branch of the portal vein
* Child-Pugh class A or B
* Performance status: ECOG 0-2 (WHO)
* Target liver lesion measurable as per WHO modified EASL criteria
* Life expectancy of at least 3 months in absence of treatments.
* Prior surgical or locoregional ablation or TACE treatments are allowed for lesions other than the target lesion treated and monitored to define tumor response.
* The following laboratory parameters must be met:

Creatinine ≤ 1.50 mg/dL, Bilirubin ≤ 2.5 mg/dL, Albumin >= 30 g/L White blood cells >= 1.5 x 109/L, PLT >= 50 x 109/L, PT >= 50%

* Signature of informed consent obtained.

Exclusion Criteria:

* Infiltrative HCC
* Liver tumor is undefined, unmeasurable or not assessable
* Occlusive thrombosis of the common portal trunk or of a main branch (right or left).
* Ascites, F3-type varices.
* Contraindications to arteriography
* Hepatofugal portal flow
* Presence of hemodynamically relevant abnormalities of hepatic arterial structure, such as not to allow for a correct and safe delivery of microspheres.
* Prior TACE to the target lesions
* Presence of chronic or acute co-morbidities (to lungs, heart, kidneys or brain) because of which the patient is not eligible to receive the treatment foreseen by the protocol.
* Prior neoplasias in the 5 preceding years or concomitance of other neoplasias at enrolment, wtih the exception of cutaneous basal cell or squamous cells carcinoma or carcinoma in situ of the uterine cervix
* Presence of localized or systemic infections (with the exception of HIV infecton responsive to therapy).
* Pregnant women (women of child-bearing potential will have a pregnancy test done) and breastfeeding women;
* Known or suspect hypersensitivity to the investigational drug or to the investigational pharmacological class;
* Patients presenting with severe clinical conditions which in the opinion of the investigator contraindicate patient participation in the study;
* Use of investigational drugs in the last month prior to inclusion into the study
* Patients who are not capable of complying with the procedures established by the protocol and of signing the informed consent. In case of minors or incapacitated patients unable to release their informed consent to take part in the study, the consent must be released and signed also by the parents/guardian or by the legal representative. Minors or incapacitated patients must as well sign the informed consent to the best of their ability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
survival of all randomized patients at month 24 (favorable event). Mortality by month 24 and withdrawal from the study will be considered to be unfavorable events. | From first TACE treatment to month 24

SECONDARY OUTCOMES:
Radiological tumor response; TTSP; TTP; Overall duration of response; Quality of life; ECOG score; Impact on liver function; No.of treatments administered. | From first TACE to month 24

CONTACTS AND LOCATIONS:
Overall Officials: Rita Golfieri, MD, Principal Investigator — Azienda Ospedaliero-Universitaria, Policlinico S.Orsola-Malpighi
Locations (5):
- Italy (5):
  - Ospedali Riuniti di Bergamo, Bergamo, BG
  - Azienda Ospedaliero-Universitaria, Policlinico S.Orsola-Malpighi, Bologna, Bologna
  - Azienda Ospedaliera Universitaria Pisana - Stabilimento di Cisanello, Pisa, PI
  - Azienda Ospadaliera Universitaria S.Giovanni Battista - Molinette, Torino, TO
  - Azienda Ospedaliera Universitaria S.Maria della Misericordia, Udine, UD